CLINICAL TRIAL: NCT05014061
Title: Adenosine's Effect on STunning Resolution in Acute Myocardial Infarction An Open-label, Single Center Trial
Brief Title: Adenosine's Effect on STunning Resolution in Acute Myocardial Infarction
Acronym: A-STAMI
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Never started
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EudraCT number: 2021-001466-37
Record Dates: First submitted 2021-07-08; First posted 2021-08-20 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2021-07

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia | interventions — Adenosine

STUDY DESIGN:
Intervention Model Description: Single center, open-label, randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adenosine (Experimental): Adenosine infusion 70 µg/kg/min initiated prior to revascularization and maintained for 6 hours
  Interventions: Drug: Adenosine
- Controll (No Intervention): Standard of care

INTERVENTIONS:
Drug: Adenosine — Adenosine infusion 70 µg/kg/min for 6 hours
  Arms: Adenosine

SUMMARY:
The aim of this study is to evaluate the effect of adenosine on the recovery of myocardial akinesia in ST-elevation myocardial infarction (STEMI). The study is a single-center randomized clinical trial intending to include 90 patients.

The objective of the study is to investigate whether treatment with adenosine hastens recovery of myocardial akinesia and improves cardiac function at 48 hours in patients with STEMI.

DETAILED DESCRIPTION:
Primary endpoint (variable):

The resolution of myocardial stunning at 48 hours (StunningRes48h).

The proportion of stunning that has resolved at 48 hours will be calculated according to the formula:

StunningRes48h = (%AkinesiaBaseline - %Akinesia48h) / (%AkinesiaBaseline - %Akinesia30days) where %AkinesiaT is defined as the endocardial length of the akinetic myocardium measured in end-diastole divided by the total endocardial length measured in end-diastole in the 2- and 4-chamber view, at time T (T= 48h or 30 days)

Secondary endpoint(s) (variables):

1. Infarct size at 6 months, as assessed by cardiac magnetic resonance imaging (magnetic resonance imaging).
2. Ejection fraction days 1, 2, 3, 7, 14, 30 and 6 months.
3. Any sustained ventricular tachycardia or fibrillation within 72 hours (safety endpoint; binary)
4. Any high-grade atrioventricular block or sinus arrest within 72 hours (safety endpoint; binary)
5. Implantation of cardiac assist device within 72 hours (binary)
6. Stroke within 6 months (binary)
7. All-cause mortality within 6 months
8. Heart failure rehospitalization within 6 months*
9. Worsening in-hospital heart failure ≥12 hours after PCI#
10. Composite of any worsening in-hospital heart failure ≥12 hours after PCI or heart failure rehospitalization within 6 months.

    * Defined as re-admission to hospital after discharge, with a total length of admission ≥24 hours, documented worsening of heart failure signs or symptoms (e.g. worsening dyspnea, fatigue, edema/fluid overload, pulmonary venous distension or signs of pulmonary edema on X-ray), with administration of intravenous diuretic or inotropic drugs, ultrafiltration, non-invasive ventilation or mechanical assist device.

      * Defined as intensification of heart failure therapy due to worsening heart failure signs or symptoms (as above; including intravenous diuretic, inotropic or vasopressor drugs, non-invasive ventilation or mechanical assist device).

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years.
2. Anterior STEMI.
3. Symptom duration ≤6 hours
4. Written informed consent obtained - Angiographic Inclusion criteria:

   1. Culprit lesion in LAD, major branch of LAD, proximal or mid LCx or proximal or mid RCA
   2. TIMI flow ≤2 in the culprit vessel

      -Echocardiographic inclusion criteria:
   3. Detectable hypo- or akinesia corresponding to ≥5% of the left ventricle corresponding to culprit lesion, per bedside visual assessment.

Exclusion Criteria:

1. Previous randomization in the study
2. Any of the following contraindications for treatment with adenosine:

   1. Known pre-existing atrioventricular block grade ≥2 or sick sinus syndrome in patients without pacemaker.
   2. Known pre-existing elevation of intracranial pressure
   3. Treatment with dipyridamole within 24 hours of randomization
   4. Systolic blood pressure <80 mm Hg at screening
3. Any concomitant condition resulting in a life expectancy of less than one month
4. Previous myocardial infarction or other cardiac condition resulting in impaired regional or global systolic function without documented recovery of cardiac function
5. Heart transplant or left ventricular assist device recipient
6. Not suitable in the opinion of the investigator due to severe or terminal comorbidity with poor prognosis or characteristics that may interfere with adherence to the trial protocol
7. Pregnancy or woman of childbearing potential who is not sterilized or using a medically accepted form of contraception -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The resolution of myocardial stunning at 48 hours (StunningRes48h). | 48 hours
  The proportion of stunning that has resolved at 48 hours will be calculated according to the formula:
  StunningRes48h = (%AkinesiaBaseline - %Akinesia48h) / (%AkinesiaBaseline - %Akinesia30days) where %AkinesiaT is defined as the endocardial length of the akinetic myocardium measured in end-diastole divided by the total endocardial length measured in end-diastole in the 2- and 4-chamber view, at time T (T= 48h or 30 days)

SECONDARY OUTCOMES:
Infarct size | 6 months
  Infarct size, assessed by cardiac magnetic resonance imaging
Ejection fraction | Day 1, Day 2, Day 3, Day 7, Day 14, Day 30 and 6 months
  Ejection fraction, assessed by echocardiography
Sustained ventricular tachycardia or fibrillation | 72 hours
  Any sustained ventricular tachycardia or fibrillation within 72 hours
High-grade atrioventricular block or sinus arrest | 72 hours
  Any high-grade atrioventricular block or sinus arrest within 72 hours
Cardiac assist device | 72 hours
  Implantation of cardiac assist device within 72 hours
Stroke | 6 months
  Stroke within 6 months
Mortality | 6 months
  All-cause mortality within 6 months
Rehospitalization | 6 months
  Heart failure rehospitalization within 6 months
Worsening heart failure | ≥12 hours
  Worsening in-hospital heart failure after PCI
Composite | ≥12 hours or 6 months
  Composite of any worsening in-hospital heart failure ≥12 hours after PCI or heart failure rehospitalization within 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Björn Redfors, MD, PhD, Principal Investigator — Vastra Gotaland Region